CLINICAL TRIAL: NCT03248934
Title: Delineating the Concurrent Validity and Diagnostic Accuracy of a Patient Performed Examination for Patients With Intra-Articular Hip Pain: A Proof of Concept Study
Brief Title: Patient Performed Examination for Patients With Intra-articular Hip Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00082395
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-05

CONDITIONS: Hip Pain Chronic; Hip Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Self-Administered Exam Group (Experimental): Participants with hip pain presenting in the hip preservation clinics will be asked to complete two diagnostic exams. Participants with hip pain will first complete a patient self-administered diagnostic exam.
  Interventions: Other: Patient Self-Administered Diagnostic Exam
- Clinician-Performed Exam Group (Active Comparator): Participants with hip pain presenting in the hip preservation clinics will be asked to complete two diagnostic exams. Participants with hip pain will next complete a clinician-performed diagnostic exam.
  Interventions: Other: Clinician-Performed Diagnostic Exam

INTERVENTIONS:
Other: Patient Self-Administered Diagnostic Exam — Participants will complete a patient self-administered diagnostic exam. A physician will be available to monitor the patient and record findings but will not physically assist the participants.
  Arms: Patient Self-Administered Exam Group
Other: Clinician-Performed Diagnostic Exam — A clinician-performed diagnostic exam will be completed on the patients.
  Arms: Clinician-Performed Exam Group

SUMMARY:
The primary objective of this study is evaluate the diagnostic accuracy of a patient self-administered clinical examination of the hip compared with a traditional clinical examination (i.e. index test).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80 years
* Seeking care for hip related pain and/or clicking, catching, giving way or stiffness
* Able to sign or verbalize study consent
* No other medical conditions (e.g. gynecological or urinary pathology) that may affect study results
* English speaking

Exclusion Criteria:

* Patients with primary lumbar spine, sacro-iliac or other non-hip related pain as determined with clinical examination
* Previous hip surgery
* Previous hip injury that would normally exclude from examination as standard practice
* Unable to sign or verbalize consent
* Other non-musculoskeletal pathology that may affect study results (e.g. gynecological or urinary pathology)
* Non-English speaking

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-03-13 (Actual)

PRIMARY OUTCOMES:
Sensitivity | End of clinician examination, 20 minutes
  As measured by a questionnaire evaluating the diagnostic test's ability to identify a positive finding when the targeted diagnosis is actually present (i.e. true positive).

SECONDARY OUTCOMES:
Specificity | End of clinician examination, 20 minutes
  As measured by the discriminatory ability of the diagnostic test to identify if the disease or condition is absent when in actuality it is truly absent (i.e. true negative).
Diagnostic accuracy measure of positive likelihood ratio | End of clinician examination, 20 minutes
  As measured by sensitivity and specificity values.
Diagnostic accuracy measure of negative likelihood ratio | End of clinician examination, 20 minutes
  As measured by sensitivity and specificity values.
Diagnostic accuracy measure of post-test probabilities | End of clinician examination, 20 minutes
  As measured by analysis of the pre-test prevalence of the condition and determination of the post-test shift in probability of the condition.

CONTACTS AND LOCATIONS:
Overall Officials: Richard C. Mather, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No